CLINICAL TRIAL: NCT02172534
Title: A Randomized, Double-blind Within Dose, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of Increasing Single and Multiple Doses (28-day Dosing) of Tiotropium Bromide Administered Once Daily Via the Respimat® Device in Cystic Fibrosis Patients
Brief Title: Safety, Tolerability and Pharmacokinetics of Tiotropium in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.338
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

ARMS (6):
- Tiotropium bromide low (Experimental): Single dose: 2.5 µg Tiotropium
  Interventions: Drug: Tiotropium bromide low
- Tiotropium bromide medium (Experimental): Single dose: 5 µg Tiotropium
  Interventions: Drug: Tiotropium bromide medium
- Tiotropium bromide high (Experimental): Single dose: 10 µg Tiotropium
  Interventions: Drug: Tiotropium bromide high
- Tiotropium bromide low (28 days) (Experimental): multiple dose: 2.5 µg Tiotropium
  Interventions: Drug: Tiotropium bromide low
- Tiotropium bromide medium (28 days) (Experimental): Multiple dose: 5 µg Tiotropium
  Interventions: Drug: Tiotropium bromide medium
- Placebo (Placebo Comparator): single or multiple dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium bromide low
  Arms: Tiotropium bromide low; Tiotropium bromide low (28 days)
Drug: Tiotropium bromide medium
  Arms: Tiotropium bromide medium; Tiotropium bromide medium (28 days)
Drug: Tiotropium bromide high
  Arms: Tiotropium bromide high
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to obtain information about the safety and tolerability of tiotropium bromide administered via the Respimat® inhalation device in pediatric (≤11 y.o.) and adolescent/adult (≥12 y.o.) cystic fibrosis (CF) patients after single and multiple doses as well as to obtain pharmacokinetic data for tiotropium in CF patients after single and multiple doses

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (pediatric ≤11 years; adolescent / adult ≥12 years)
* Documented diagnosis of CF (positive sweat chloride ≥60 mEq/liter, by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF accompanied by one or more clinical features with the CF phenotype
* Able to perform acceptable spirometric maneuvers, according to ATS (American Thoracic Society) standards
* FEV1 >25% of predicted values
* Patients must be able to inhale medication in a reproducible manner from the Respimat® inhaler and from a metered dose inhaler (MDI)
* Clinical stability:

  * no evidence of acute upper or lower respiratory tract infection within 4 weeks of screening
  * no pulmonary exacerbation requiring use of i.v./oral/inhaled antibiotics, or oral corticosteroids within 4 weeks of screening
  * FEV1 at Visit 2 must be within 10% of FEV1 at Visit 1. If FEV1 at Visit 2 is not within 10% of FEV1 at Visit 1, Visit 2 may be re-scheduled once within 7 days
* The patient or the patient's legally acceptable representative must be able to give informed consent in accordance with International Conference on Harmonization (ICH) Good Clinical Practice (GCP) guidelines and local regulation
* Patients taking a chronic medication must be willing to continue this therapy for the entire duration of the study

Exclusion Criteria:

* Patients with a significant history of allergy / hypersensitivity (including medication allergy) which is deemed relevant to the trial as judged by the Investigator. "Relevance" in this context refers to any increased risk of hypersensitivity reaction to trial medication
* Patients with a known hypersensitivity to study drug or its components
* Patients who have participated in another study with an Investigational drug within one month or six half-lives (whichever is greater) preceding the screening visit
* Patients who are currently participating in another trial. Observational studies are allowed. Permission should be obtained from the sponsor of the study
* Patients with known relevant substance abuse, including alcohol or drug abuse. The intention of this criterion was to exclude patients who are considered to be at risk of not complying with or abusing the trial medication administration directives.
* Female patients who are pregnant or lactating, including females who have a positive urine pregnancy test at screening (pregnancy tests were performed for all females of child bearing potential)
* Female patients of child bearing potential who are not using a medically approved form of contraception.
* Patients with documented persistent colonization with B. cepacia (defined as more than one positive culture within the past year). The intention of this exclusion criterion is to be consistent with the current policy within the CF community for reducing the risk of B. cepacia cross infection.
* Patients who have started a new chronic medication for CF within four (4) weeks of screening. Patients who are on a cycling TOBI® (Tobramycin treatment) regimen must have completed at least three (3) cycles of every other month TOBI® administration prior to the screening visit. As there are other cycles used with TOBI®, the clinical monitor should be consulted before the patient was enrolled.
* Clinically significant disease or medical condition other than CF or CF-related conditions that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data. This included significant hematological, hepatic, renal, cardiovascular, and neurologic disease. Patients with diabetes could participate if their disease is under good control prior to screening. This criterion provides an opportunity for the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in physical examination | Baseline, Day 1 and 28
Changes from baseline in blood pressure | Baseline, Day 1 and 28
Changes from baseline in pulse rate | Baseline, Day 1 and 28
Changes from baseline in laboratory evaluation | Baseline, Day 28
Occurrence of Adverse Events | up to 59 days
Change in FEV1 (Forced expiratory volume in one second) | Pre-dose and 0.5, 1 and 2 hours after treatment on Day1 and 28
Change in FVC (Forced vital capacity) | Pre-dose and 0.5, 1 and 2 hours after treatment on Day1 and 28
Change in FEF25-75% (Forced Expiratory Flow) | Pre-dose and 0.5, 1 and 2 hours after treatment on Day1 and 28

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) after the first dose of 2.5 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
tmax (time from dosing to maximum concentration) after the first dose of 2.5 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point within the first dosing of 2.5 μg tiotropium bromide interval) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) after the first dose of 2.5 μg tiotropium bromide | Pre-dose and 0-2, 2-4 and 4-8 hours after treatment on Day1
fet1-t2 (fraction of analyte excreted in urine from time point t1 to t2) after the first dose of 2.5 μg tiotropium bromide | Pre-dose and 0-2, 2-4 and 4-8 hours after treatment on Day1
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
%AUCtz-∞ (the percentage of the AUC 0-∞ that is obtained by extrapolation) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
λz (terminal rate constant of the analyte in plasma) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
t½ (terminal half-life of the analyte in plasma) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
MRTih (mean residence time of the analyte in the body after inhalation) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
Vz/F (apparent volume of distribution of the analyte during the terminal phase λz following an extravascular dose) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
CLR,t1- t2 (renal clearance of the analyte in plasma from the time point t1 to time point t2) after the first dose of 5 μg and 10 μg tiotropium bromide | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day1
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
Cpre,ss(predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
λz,ss (terminal rate constant in plasma at steady state) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
MRTih,ss (mean residence time of the analyte in the body after 14 administrations at steady state) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
CL/F,ss (apparent clearance of the analyte in the plasma at steady state following extravascular multiple dose administration) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
Aet1-t2,ss (amount of analyte that is eliminated in urine at steady state from the time point t1 to time point t2) | Pre-dose and 0-2, 2-4 and 4-8 hours after treatment on Day 28
fet1-t2,ss (fraction of analyte eliminated in urine at steady state from time point t1 to time point t2) | Pre-dose and 0-2, 2-4 and 4-8 hours after treatment on Day 28
CLR,t1-t2,ss (renal clearance of the analyte in plasma from the time point t1 until the time point t2 at steady state) | Pre-dose and 5, 15, 30 min and 1, 2, 4, 6 hours after treatment on Day 28
Accumulation Ratio (R)A,Cmax,28 based on Cmax | 28 days
Accumulation Ratio (R)A,AUC,28 based on AUC0-τ | 28 days
Linearity index (LI) | 28 days